CLINICAL TRIAL: NCT01537510
Title: Accelerating Adoption of Childhood Obesity Comparative Effectiveness Research
Brief Title: Study of Technology to Accelerate Research
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Brigham and Women's Hospital (Other); Cambridge Health Alliance (Other); Harvard Vanguard Medical Associates (Other)
Responsible Party: Principal Investigator, Elsie Taveras, Associate Professor of Population Medicine, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R18AE000026 (NIH)
Record Dates: First submitted 2012-02-07; First posted 2012-02-23 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Usual Care (Active Comparator)
  Interventions: Behavioral: STAR - Study of Technology to Accelerate Research
- Clinician intervention only (Experimental): This arm will entail the development and deployment of alerts and access to a SmartSet at the time of a well child visit with a child between the ages of 6-12 years with a BMI ≥ 95th percentile.
  Interventions: Behavioral: STAR - Study of Technology to Accelerate Research
- Clinician intervention plus Direct-to-parent communication (Experimental): Parents of children enrolled in this intervention arm will receive mailings, text messages and a series of 4 calls with a health coach to encourage behavior change in addition to the intervention received by the clinicians.
  Interventions: Behavioral: STAR - Study of Technology to Accelerate Research

INTERVENTIONS:
Behavioral: STAR - Study of Technology to Accelerate Research — In 14 pediatric practices, to conduct a cluster-randomized controlled trial to examine the extent to which computerized point of care decision alerts to pediatric primary care providers, with or without direct-to-parent communications, will increase adoption of comparative effectiveness research evidence on childhood obesity for children 6 to 12 years of age with a BMI ≥ 95th percentile.

SUMMARY:
Childhood obesity is highly prevalent and is associated with both short- and long-term adverse outcomes.

Despite availability of guidelines for nearly a decade and more recent comparative effectiveness research (CER) evidence, the health care system has been slow to adopt recommended practices. Although pediatric health care providers often cite barriers such as limited time, skill, and resources, a frequently overlooked barrier is the lack of data systems to efficiently and accurately assess guideline implementation and to improve quality of care for childhood obesity. Health information technology (HIT) offers potential for accelerating the adoption of CER evidence regarding childhood obesity screening and management, for establishing treatment benchmarks, and for supporting patients and their clinical teams in care improvement. Incorporation of HIT may be especially effective if augmented by outreach to parents and children.

The goal of this study is to develop and test system-level interventions to accelerate the adoption of CER evidence on childhood obesity screening and management, and ultimately improve obesity-related health care quality and outcomes. To achieve this goal, the investigators will work with two health care systems in Massachusetts with strong track records of research collaboration: Cambridge Health Alliance (CHA), an integrated academic public health system, and Harvard Vanguard Medical Associates (HVMA), a large multi-site group practice. Both systems use an electronic medical record for all aspects of ambulatory care, including point of care services such as electronic order entry and centralized functions such as patient scheduling.

In these settings of innovation and commitment to improving quality of care, the investigators will develop and test two systematic strategies for adoption of CER evidence. The first incorporates computerized point of care decision alerts to pediatric primary care providers during routine office visits, linked to CER-based algorithms of care. The second augments this HIT approach with direct-to-parent communication of child's body mass index (BMI) along with recommended evaluation and management. The specific aims of this study are:

1. In 18 community health centers of CHA, to identify barriers to and facilitators of adoption of an existing set of computerized point of care decision alerts for childhood obesity screening and management. The investigators will achieve this aim through in-depth interviews and surveys with primary care clinicians, which will inform the design of the investigators proposed intervention.
2. In 14 practices of HVMA, to conduct a cluster-randomized controlled trial to examine the extent to which computerized point of care decision alerts to pediatric primary care providers, with or without direct-to-parent communications, will increase adoption of CER evidence on childhood obesity for children 6 to 12 years of age with a BMI ≥ 95th percentile. The investigators will determine the extent to which each of the 2 intervention conditions, compared with the usual care control condition and with each other, results in:

   1. Increased screening and assessment of childhood obesity at the point of care, including BMI, blood pressure, and laboratory screening, and provision of nutrition and physical activity counseling,
   2. A smaller age-associated increase in BMI over a 1-year period, and,
   3. Improved specific dietary, physical activity, and sedentary behaviors over a 1-year period.
3. To evaluate each intervention's costs (including clinician and family time) and cost-effectiveness in terms of children's change in BMI and weight-related behaviors.
4. To develop a detailed dissemination guide to further accelerate adoption of CER evidence on childhood obesity in practices and communities interested in implementing similar interventions.

To achieve the investigators aims, the investigators have assembled a research team with extensive experience in obesity prevention, clinician and child behavior change, clinical informatics, statistical methodology in cluster randomized controlled trials, cost-effectiveness analyses, and dissemination science. If successful, this project will provide new and sustainable approaches for accelerating adoption of CER evidence for childhood obesity screening and management and for improving quality of care for childhood obesity in pediatric primary care.

ELIGIBILITY:
Inclusion Criteria:

* child is age 6.0 through 12.9 years at baseline
* child's BMI exceeds the 95th percentile for age and sex (CDC criteria
* parent can respond to interviews and questionnaires in English
* child has obtained well-child care from HVMA for at least the previous 15 months.

Exclusion Criteria:

* children who do not have at least one parent who is able to follow study procedures for 1 year
* families who plan to leave HVMA within the study time frame
* families for whom the primary care clinician thinks the intervention is inappropriate, e.g., emotional or mental difficulties
* children with chronic conditions that substantially interfere with growth

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 549 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in screening and assessment of childhood obesity at the point of care, including BMI, blood pressure, and laboratory screening, and provision of nutrition and physical activity counseling | Baseline and 1 Year

SECONDARY OUTCOMES:
Change in Body Mass Index | Baseline and 1 year
  Outcomes at 1 year will include changes from baseline in Body mass index defined as the ratio of weight (kg) to the square of standing height (m)
Change in Health Behaviors | Baseline and 1 year
  1) Sugar-sweetened beverage intake, 2) Fast food, 3) Physical activity, 4) TV viewing and 5) sleep.
Costs (including clinician and family time) and cost-effectiveness in terms of children's change in BMI and weight-related behaviors | For the duration of the intervention, from planning through completion of the intervention, up to 3 years
  We will study the costs of our intervention with two goals: (a) to inform clinicians and policymakers about what investment would be required to adopt this intervention in other settings, and (b) to generate key assumptions for analysis of the cost-effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Elsie M Taveras, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care Institute/Harvard Medical School
Locations (1):
- Harvard Vanguard Medical Associates, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fiechtner L, Fonte ML, Castro I, Gerber M, Horan C, Sharifi M, Cena H, Taveras EM. Determinants of Binge Eating Symptoms in Children with Overweight/Obesity. Child Obes. 2018 Nov/Dec;14(8):510-517. doi: 10.1089/chi.2017.0311. Epub 2018 Aug 28. PMID 30153037
- [Derived] Taveras EM, Marshall R, Kleinman KP, Gillman MW, Hacker K, Horan CM, Smith RL, Price S, Sharifi M, Rifas-Shiman SL, Simon SR. Comparative effectiveness of childhood obesity interventions in pediatric primary care: a cluster-randomized clinical trial. JAMA Pediatr. 2015 Jun;169(6):535-42. doi: 10.1001/jamapediatrics.2015.0182. PMID 25895016
- [Derived] Taveras EM, Marshall R, Horan CM, Gillman MW, Hacker K, Kleinman KP, Koziol R, Price S, Simon SR. Rationale and design of the STAR randomized controlled trial to accelerate adoption of childhood obesity comparative effectiveness research. Contemp Clin Trials. 2013 Jan;34(1):101-8. doi: 10.1016/j.cct.2012.10.005. Epub 2012 Oct 22. PMID 23099100